CLINICAL TRIAL: NCT02059083
Title: Biofeedback for Adolescent Cannabis Use Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding not received; study was never started
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0412
Record Dates: First submitted 2014-02-05; First posted 2014-02-11 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Adolescent Cannabis Use Disorder
Keywords: adolescent; cannabis; biofeedback
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (CBT) alone (Active Comparator)
  Interventions: Behavioral: CBT
- Cognitive behavioral therapy plus HRV biofeedback (Experimental)
  Interventions: Behavioral: Heart rate variability biofeedback

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback
  Arms: Cognitive behavioral therapy plus HRV biofeedback
Behavioral: CBT
  Arms: Cognitive behavioral therapy (CBT) alone

SUMMARY:
The aims of this study are: 1) to estimate the effect size of HRV biofeedback for stress in adolescents undergoing cognitive behavioral therapy (CBT) for cannabis use disorder (primary outcome: Perceived Stress Scale) and 2) to estimate the effect size of HRV biofeedback for cannabis use in adolescents undergoing CBT for cannabis use disorder (primary outcome: number of days used cannabis in the past 30 days).

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 13 and 19 years, with a parent or legal guardian available to complete parental assessments, if the participant is a minor
* meet Diagnostic and Statistical Manual of Mental Disorders, 5th edition, (DSM-V) criteria for cannabis use disorder by clinical interview;
* be medically healthy;
* be willing to participate in the study intervention and assessments;
* plan to live locally for at least 4 months;
* be able to read English well enough to complete study questionnaires;
* have self-reported cannabis use in the past 28 days;
* have a Perceived Stress Scale score > 20.

Exclusion Criteria:

* current or past psychosis;
* bipolar I or II disorder;
* the need to take psychotropic medications at any time during the study;
* pregnancy;
* psychiatric or substance use disorder that cannot be managed with outpatient care (e.g. alcohol withdrawal, severe major depressive disorder, significant suicidal ideation); and
* medications known to affect HRV (e.g. albuterol, pseudoephedrine, beta adrenergic blockers).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale | baseline and 16 weeks

SECONDARY OUTCOMES:
Change in the number of days used marijuana in the past 28 days | baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Thurstone, M.D., Principal Investigator — Denver Health